CLINICAL TRIAL: NCT07319546
Title: Effectiveness of Accelerated Rehabilitation on Knee Joint Function and Quality of Life in Individuals With Total Knee Arthroplasty: A Double Blind Randomized Controlled Trial
Brief Title: Accelerated Rehabilitation in Individuals After Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2025/443.2908
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthristis; Arthroplasties, Knee Replacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated rehabilitation (Experimental): Rehabilitaion after TKR with the accelerated and optimal loading concepts
  Interventions: Behavioral: Accelerated exercise
- Conventional rehabilitation (Active Comparator)
  Interventions: Behavioral: Routine exercise

INTERVENTIONS:
Behavioral: Accelerated exercise — Based on optimal and accelerated concepts
  Arms: Accelerated rehabilitation
Behavioral: Routine exercise — Conventional program
  Arms: Conventional rehabilitation

SUMMARY:
The primary aim of this double-blind randomized controlled trial is to evaluate the effectiveness of an accelerated rehabilitation protocol on knee joint function and quality of life in individuals undergoing TKA compared to conventional rehabilitation in Dali, Yunan, China. The study will include patients aged 50-80 years who are scheduled for primary unilateral TKA. Participants will be randomly assigned to either an accelerated rehabilitation group or conventional rehabilitation group. The primary outcomes will include knee joint function, assessed using the KOOS and quality of life measures using the SF-36 surveys. The study will follow participants for 6 months post-surgery to assess longer-term outcomes. This study will not include individuals undergoing revision TKA or those with severe comorbid conditions. The results will provide critical insights into the role of accelerated rehabilitation in improving post-operative recovery, functional outcomes, and overall quality of life for TKA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with end-stage knee OA necessitating primary unilateral TKA.

Exclusion Criteria:

* History of joint infections, cancer, or inflammatory arthritis.
* End-stage OA from rheumatoid or septic arthritis.
* Individuals with neurological disorders such as Alzheimer's disease, - Parkinson's disease, stroke.
* Individuals who are unable to follow a structured rehabilitation protocol.
* Previous history of knee surgeries (other than arthroscopy).
* Severe comorbidities that would hinder participation (e.g., advanced cardiovascular diseases).
* Individuals who have severe osteoporosis.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | From enrollment to the end of 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Komsak Sinsurin, Ph.D., DPT, Study Chair — Mahidol University; Liying Yang, Principal Investigator — West Yunnan University of Applied Sciences, Yunnan province
Locations (1):
- Hospital, Dali, Yunnan, China

IPD SHARING:
Plan to Share IPD: No